CLINICAL TRIAL: NCT00006294
Title: Pharmacological Association of the Angiotensin-Converting Enzyme Insertion/Deletion Polymorphism on Blood Pressure and Cardiovascular Risk in Relation to Anti-hypertensive Treatment
Brief Title: Genetics of Hypertension Associated Treatments (GenHAT)
Acronym: GenHAT
Status: Completed | Type: Observational
Sponsor: Donna Arnett, 257-5678 (Other)
Collaborators: University of Minnesota (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Donna Arnett, 257-5678, PI, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 911; R01HL063082 (NIH)
Record Dates: First submitted 2000-09-25; First posted 2000-09-26 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Coronary Disease; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Coronary Disease; Myocardial Infarction | interventions — Chlorthalidone; Lisinopril; hydrochlorothiazide, lisinopril drug combination; Amlodipine; Doxazosin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chlorthalidone: Participants will take chlorthalidone at recommended doses to control hypertension
  Interventions: Drug: Chlorthalidone
- Amlodipine: Participants will take Amlodipine at recommended doses to control hypertension
  Interventions: Drug: Amlodipine
- Lisinopril: Participants will take Lisinopril at recommended doses to control hypertension
  Interventions: Drug: Lisinopril
- Doxazosin: Participants will take Doxazosin at recommended doses to control hypertension
  Interventions: Drug: Doxazosin

INTERVENTIONS:
Drug: Chlorthalidone — participant's drug dose will be titrated from 12.5mg to 25mg over the course of the study
  Other Names: Hygroton, Thalitone, Chlorthalid
  Groups: Chlorthalidone
Drug: Lisinopril — participant's drug dose will be titrated from 10mg to 40mg over the course of the study
  Other Names: Zestoretic
  Groups: Lisinopril
Drug: Amlodipine — participant's drug dose will be titrated from 10mg to 40mg over the course of the study
  Other Names: Norvasc
  Groups: Amlodipine
Drug: Doxazosin — participant's drug dose will be titrated from 2mg to 8mg over the course of the study
  Other Names: Cardura
  Groups: Doxazosin

SUMMARY:
To examine whether the association between selected hypertensive genes and combined fatal coronary heart disease and nonfatal myocardial infarction in high-risk hypertensives is modified by the type of antihypertensive treatment, leading to differential risks of coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

The study might shed important light on the variation in patient response to antihypertensive agents, and improve the ability to pick the right antihypertensive for specific patients. GenHAT is an ancillary study to ALLHAT (the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial). ALLHAT recruited 42,515 hypertensives and randomized them to one of four antihypertensive agents (lisinopril, chlorthalidone, amlodipine, and doxazosin); follow-up will be completed in March, 2002.

DESIGN NARRATIVE:

GenHAT, a prospective study ancillary to ALLHAT, will characterize hypertension genetic variants and determine their interaction with antihypertensive treatments in relation to coronary heart disease (CHD). DNA from frozen clots stored at the ALLHAT Central Laboratory will be used to genotype variants of hypertension genes (angiotensinogen -6, angiotensin converting enzyme insertion/deletion, angiotensin type- 1 receptor, alpha-adducin, beta2 adrenergic receptor, lipoprotein lipase, and 10 new hypertension variants expected to be discovered during the course of the study). In addition to the primary aim, a number of secondary aims will be undertaken to evaluate gene- treatment interactions in relation to other endpoints, including all-cause mortality, stroke, heart failure, left ventricular hypertrophy, decreased renal function, peripheral arterial disease, and blood pressure lowering. Because of the ethnic and gender diversity of ALLHAT, an assessment will be made of the effects of these variants on outcomes in key subgroups (age >65 years, women, African Americans, Type II diabetics), and whether the gene-treatment interactions in relation to outcomes are consistent across subgroups.

ELIGIBILITY:
* not taking anti-hypertensive medication
* use of anti-hypertensives for less than two months with a baseline blood pressure between 140/90 and 180/110
* use of anti-hypertensives for greater than two months with a blood pressure not greater than 160/100
* at least one additional cardiovascular risk factor such as previous MI, stroke, type 2 diabetes, smoking, left ventricular hypertrophy or dyslipidemia

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive individuals, multiple races and ethnic groups are represented in this study population
Sampling Method: Probability Sample
Enrollment: 37939 (Actual)
Dates: Start 1999-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | baseline and six month
  Blood pressure will be measured to determine the effect of the prescribed anti-hypertensive . Data will be presented as the change in blood pressure over the course of six months

SECONDARY OUTCOMES:
Effect of genotype on event rates | 6 years
  The rate of fatal myocardial infarction (MI) was evaluated in relation to the ACE I/D genotype and anti-hypertensive used. Data are presented as the incidence of fatal MI after six years of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Donna Arnett, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Background] Arnett DK, Boerwinkle E, Davis BR, Eckfeldt J, Ford CE, Black H. Pharmacogenetic approaches to hypertension therapy: design and rationale for the Genetics of Hypertension Associated Treatment (GenHAT) study. Pharmacogenomics J. 2002;2(5):309-17. doi: 10.1038/sj.tpj.6500113. PMID 12439737
- [Background] Arnett DK, Davis BR, Ford CE, Boerwinkle E, Leiendecker-Foster C, Miller MB, Black H, Eckfeldt JH. Pharmacogenetic association of the angiotensin-converting enzyme insertion/deletion polymorphism on blood pressure and cardiovascular risk in relation to antihypertensive treatment: the Genetics of Hypertension-Associated Treatment (GenHAT) study. Circulation. 2005 Jun 28;111(25):3374-83. doi: 10.1161/CIRCULATIONAHA.104.504639. Epub 2005 Jun 20. PMID 15967849
- [Derived] Zhang X, Lynch AI, Davis BR, Ford CE, Boerwinkle E, Eckfeldt JH, Leiendecker-Foster C, Arnett DK. Pharmacogenetic association of NOS3 variants with cardiovascular disease in patients with hypertension: the GenHAT study. PLoS One. 2012;7(3):e34217. doi: 10.1371/journal.pone.0034217. Epub 2012 Mar 28. PMID 22470539